CLINICAL TRIAL: NCT00119717
Title: Safety and Efficacy of NeuroFlo Technology in Ischemic Stroke (SENTIS)
Acronym: SENTIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CoAxia (Industry)
Responsible Party: Ashfaq Shuaib, MD, University of Alberta, Edmonton
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CD-0125
Record Dates: First submitted 2005-07-07; First posted 2005-07-14 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Cerebrovascular Accident
Keywords: acute; ischemic; stroke; randomized; device; treatment
MeSH Terms: conditions — Stroke; Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Device: NeuroFlo™ catheter
- 2 (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Device: NeuroFlo™ catheter — 45 minute treatment
  Arms: 1
Other: Control — ASA Guidelines
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the NeuroFlo™ catheter for use in patients with ischemic stroke. The NeuroFlo device is intended to increase blood flow to the brain and potentially reduce the damage caused by stroke.

DETAILED DESCRIPTION:
The study is a prospective, controlled, randomized, single-blind, multi-center study of NeuroFlo treatment plus standard medical management versus standard medical management alone. Randomization will be 1:1 and stratified to ensure equivalent patient distribution between treatment and control for the following key parameters:

1. National Institute of Health Stroke Scale (NIHSS) at baseline (stratify <10, 11-18)
2. Time from symptom onset (TFSO) to time of baseline NIHSS evaluation (stratify <5 hrs, or ≥5 hrs).

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke
* NIHSS between 5-18
* Time from symptom onset less than 14 hours

Exclusion Criteria:

* Hemorrhagic stroke
* Certain types of heart disease
* Kidney disease
* Other conditions the doctor will assess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2005-06; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The safety of the NeuroFlo device and procedure will be compared to medical management alone | 90 days
Efficacy will be assessed using a global outcome score | 90 days

SECONDARY OUTCOMES:
Acute improvement in neurological function | 24 hours
Stroke Impact Scale | 30 & 90 days
Hospital length of stay | Varies
Patient disposition upon discharge will be compared | Varies

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Shuaib, MD, Principal Investigator — University of Alberta, Edmonton
Locations (72):
- United States (47):
  - Huntsville Hospital, Huntsville, Alabama
  - UCLA, Los Angeles, California
  - Good Samaritan Hospital, San Jose, California
  - Morton Plant Hospital, Clearwater, Florida
  - University of Florida, Jacksonville, Florida
  - Univ. of Miami, Miami, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - The Queen's Medical Center, Honolulu, Hawaii
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Michigan State University, Lansing, Michigan
  - St. Joseph Mercy - Oakland, Pontiac, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Providence Hospital, Southfield, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Sunrise Medical Center, Las Vegas, Nevada
  - JFK Medical Center, Edison, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - SUNY-Upstate Medical Univ., Syracuse, New York
  - Univeristy of North Carolina, Chapel Hill, North Carolina
  - Presbyterian Hospital, Charlotte, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Sacred Heart Medical Center, Springfield, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - St. Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Brackenridge Hospital/Seton Medical Center, Austin, Texas
  - Methodist Hospital, Houston, Texas
  - Neurological Associates/CJW Med Ctr, Richmond, Virginia
  - Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Austria (3):
  - AKH General Hospital, Linz
  - Christian-Doppler-Klinik, Salzburg
  - Donauklinikum Tulln, Tulln
- Belgium (3):
  - ZNA Middelheim, Antwerp
  - AZ St Jan Brugge, Bruges
  - UZ Gasthuisberg, Leuven
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Western Ontario, London, Ontario
  - Trillium Health Centre, Mississauga, Ontario
- Germany (6):
  - Klinikum Köln-Merheim, Cologne
  - Universitatsklinikum Erlangen, Erlangen
  - Universitatsklinikum Duisberg-Essen, Essen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitatsklinikum Mannheim, Mannheim
  - Dr. Horst Schmidt Kliniken, Wiesbaden
- Medical Health and Science Center, University Of Debrecen, Debrecen, Hungary
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Hebrew University, Jerusalem
  - Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- University of Puerto Rico, San Juan, Puerto Rico
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
- Switzerland (2):
  - InselSpital, Bern
  - CHUV, Lausanne

REFERENCES:
- [Result] Shuaib A, Bornstein NM, Diener HC, Dillon W, Fisher M, Hammer MD, Molina CA, Rutledge JN, Saver JL, Schellinger PD, Shownkeen H; SENTIS Trial Investigators. Partial aortic occlusion for cerebral perfusion augmentation: safety and efficacy of NeuroFlo in Acute Ischemic Stroke trial. Stroke. 2011 Jun;42(6):1680-90. doi: 10.1161/STROKEAHA.110.609933. Epub 2011 May 12. PMID 21566232
- [Derived] Schellinger PD, Shuaib A, Kohrmann M, Liebeskind DS, Jovin T, Hammer MD, Sen S, Huang DY, Solander S, Gupta R, Leker RR, Saver JL; SENTIS Trial Investigators. Reduced mortality and severe disability rates in the SENTIS trial. AJNR Am J Neuroradiol. 2013 Dec;34(12):2312-6. doi: 10.3174/ajnr.A3613. Epub 2013 Jul 4. PMID 23828106
- [Derived] Schellinger PD, Kohrmann M, Liu S, Dillon WP, Nogueira RG, Shuaib A, Liebeskind DS; SENTIS Trial Investigators. Favorable vascular profile is an independent predictor of outcome: a post hoc analysis of the safety and efficacy of NeuroFlo Technology in Ischemic Stroke trial. Stroke. 2013 Jun;44(6):1606-8. doi: 10.1161/STROKEAHA.111.000709. Epub 2013 Apr 2. PMID 23549132
- [Derived] Shuaib A, Schwab S, Rutledge JN, Starkman S, Liebeskind DS, Bernardini GL, Boulos A, Abou-Chebl A, Huang DY, Vanhooren G, Cruz-Flores S, Klucznik RP, Saver JL; SENTIS trial investigators. Importance of proper patient selection and endpoint selection in evaluation of new therapies in acute stroke: further analysis of the SENTIS trial. J Neurointerv Surg. 2013 May;5 Suppl 1(0 1):i21-4. doi: 10.1136/neurintsurg-2012-010562. Epub 2013 Jan 3. PMID 23291425
- See also: Related Info — http://www.coaxia.com